CLINICAL TRIAL: NCT04915261
Title: A Randomized Trial of Lenient Versus Strict Arm Instruction Post Cardiac Device Surgery - LENIENT
Brief Title: A Randomized Trial of Lenient Versus Strict Arm Instruction Post Cardiac Device Surgery
Acronym: LENIENT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Principal Investigator, David Birnie, Deputy Chief, Division of Cardiology, University of Ottawa Heart Institute, Ottawa Heart Institute Research Corporation
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 20210168-01H
Record Dates: First submitted 2021-05-31; First posted 2021-06-07 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Post-Op Complication
Keywords: Cardiac; Implantable; Electronic; Device; Arm; Restriction; Post-operative; infection; dislodgement; hematoma; DVT
MeSH Terms: conditions — Postoperative Complications; Infections; Hematoma

STUDY DESIGN:
Intervention Model Description: The trial is a single centre non-inferiority cluster crossover trial. Arm restriction protocol will cross over every 8 months with a one month run-in then 7 months of data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strict Arm (Active Comparator): The strict arm group will be given the following restrictions. These restrictions are the current institutional protocol at the study site and falls within common practice pattern across Canada:
  1. No arm or shoulder movement x 24 hours
  2. No movement of affected arm overhead x 8 weeks
  3. No lifting anything heavier than 5 lbs (2.5kg) and avoid any kind of sports or other vigorous activities including golf, tennis, swimming or sweeping x 8 weeks
  4. Avoid any kind of shovelling x 8 weeks
  Interventions: Behavioral: Strict Arm Restriction
- Lenient Arm (Active Comparator): The lenient arm restriction group will be given the following restrictions. The justification for the selected lenient restriction is based on the current recommendations at a Canadian center as identified by the national survey:
  1. No shoveling 7 days,
  2. No golfing/swimming/tennis 14 days
  3. No other restrictions (overhead activity and weight lifting no limitation)
  Interventions: Behavioral: Lenient Arm Restriction

INTERVENTIONS:
Behavioral: Lenient Arm Restriction — The study will crossover between either strict arm restriction guidelines for patients or lenient arm restrictions.
  Arms: Lenient Arm
Behavioral: Strict Arm Restriction — The study will crossover between either strict arm restriction guidelines for patients or lenient arm restrictions.
  Arms: Strict Arm

SUMMARY:
The purpose and objectives of this study is to investigate whether reducing the existing arm restrictions on patients who receive Cardiac Implantable Electronic Devices (CIED) will result in an improved patient experience post operatively and reduce complication rates. There are multiple and varied arm restriction instructions given to patients receiving CIED's with limited universally accepted protocols or advice on restrictions for patients following surgery.

Restrictions such as arm immobilization, showering and weight lifting, in addition to contradictory advice between various hospitals and physicians, can negatively affect patient quality of life and increase patient anxiety with no current evidence for benefit. A cluster cross over randomized trial has been designed to test the comparative effectiveness of lenient vs strict arm restrictions for all patients receiving implantable devices.

Instructions within both arms of this study are considered within reasonable practice in Canada.

All arm restriction instructions and parameters will be embedded within EPIC, nurses will teach the restriction in addition they will be provide to the patients via printed EPIC discharge summaries. Further links will be embedded in the After Visit Summary (AFS) printouts and my Chart for patients in EPIC. These instructions will be changed every 8 months, as per the crossover design of the trial. Additionally, both arms will utilize interactive voice recognition (IVR) to provide patients with further reminders and instruction on arm restrictions.

All patients are given standard of care instructions for follow up and complication assessment through the investigators' device clinic and 24/7 on call nursing program.

DETAILED DESCRIPTION:
The purpose and objectives of this study is to investigate whether reducing the existing restrictions on patients post CIED will result in an improved patient experience post operatively and reduce complication rates. Results from this study will create standardized, postoperative arm restriction recommendations more uniform between various hospitals.

Hypothesis: The investigators hypothesize that outcomes of the post CIED implanted patients given lenient arm restriction will be non-inferior to those with prolonged arm restriction at reducing a combined primary endpoint of lead dislodgement, device infection, clinically significant pocket hematoma, upper limb DVT and frozen shoulder.

Clinical relevance: The investigators anticipate that patients with minimal (lenient) arm restriction will have similar postoperative complication rates compared to the prolonged arm restriction. Should this hypothesis be proven, this will greatly improve patient quality of life post CIED with less stringent restrictions.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing device surgery which includes implantation of at least one new endovascular lead

Exclusion Criteria:

* Standalone CIED generator replacement
* Subcutaneous implantable cardioverter defibrillators
* Leadless endocardial pacemakers
* Temporary permanent pacemakers

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6300 (Estimated)
Dates: Start 2021-08-19 (Actual); Primary Completion 2029-08-01 (Estimated); Study Completion 2030-08-01 (Estimated)

PRIMARY OUTCOMES:
A composite of 1) Lead dislodgement 2) Frozen shoulder 3) Upper arm venous thrombosis 4) Clinically significant hematoma formation | 1 year
  Definitions of each component of primary outcome:
  1. Lead dislodgement; dislodgment requiring surgical repair and dislodgement not occurring in the immediate post-op period (i.e., before the randomized intervention begins). Immediate post-op period is defined as from pocket closure to dislodgement suspected on first post- operative CXR (which is done 2-4hrs post-op).
  2. Frozen shoulder in this study is defined as: Nursing or physician note mention of chronologically related (to index surgery) patient complaint of new or markedly worsened shoulder pain and/or restricted and stiffness of active and passive range of motion.
  3. Upper arm venous thrombosis.
  4. Clinically significant hematoma is defined as done in BRUISE CONTROL 2 trial: a hematoma that required re-operation and/or resulted in prolongation of hospitalization and/or required interruption of oral anticoagulation.

SECONDARY OUTCOMES:
Rate of hematoma | 1 year
  1. Rate of hematoma (# of clinically significant hematoma / total number of procedures performed for each arm)
Rate of lead dislodgement | 1 year
  2. Rate of lead dislodgement (# of lead dislodgements / total number of new leads placed in each arm) separate by type of lead (RA vs. RV vs. LV)
Rate of frozen shoulder | 1 year
  3. Rate of frozen shoulder (# of frozen shoulders / total number of procedures performed for each arm)

CONTACTS AND LOCATIONS:
Overall Officials: David Birnie, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Golian M, Sadek MM, Aydin A, Davis D, Green M, Klein A, Nair GM, Nery P, Ramirez FD, Redpath C, Hansom SP, Wells GA, Birnie DH. A Randomized Trial of Lenient Versus Strict Arm Instruction Post Cardiac Device Surgery (LENIENT). Am Heart J. 2023 May;259:52-57. doi: 10.1016/j.ahj.2023.01.016. Epub 2023 Jan 25. PMID 36708911